CLINICAL TRIAL: NCT00435968
Title: Safety and Immune Enhancing Effects of Acute Dosing of COLD-fX in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CV Technologies (Industry)
Organization: Afexa Life Sciences Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVT-E002-2006-1
Record Dates: First submitted 2007-02-14; First posted 2007-02-16 (Estimated); Last update posted 2007-07-17 (Estimated); Status verified 2007-07

CONDITIONS: Healthy
Keywords: NK Cells; Cytokines; Lymphocytes; Immunoglobulins; Th1 response
MeSH Terms: interventions — COLD-fX

INTERVENTIONS:
Drug: CVT E002 (Cold-fX)

SUMMARY:
Subjects will be asked to participate in a four day research study of the immune system effects and safety of short-term acute dosing of Cold-fX.

The purpose of the study is to determine the effects of acute dosing of Cold-fX for 3 days on the immune system compared to a placebo (dummy pill). Safety of the acute dosing will be determined through various blood tests carried out during the study.

DETAILED DESCRIPTION:
Eligible volunteers from Hackensack University Medical Centre will be randomly assigned to either the treatment or placebo group with equal numbers in each group.

The treatment will consist of taking three capsules of CVT-E002 (600mg) or placebo three times daily on Day 1, two capsules of CVT-E002 (400mg) or placebo three times daily on Day 2 and one capsule of CVT-E002 (200mg) or placebo three times daily on Day 3.

A fasting blood sample will be collected on all 4 days of study participation. Immunological assays and blood chemisty safety tests will be performed on the samples. Serum samples will also be collected and stored until futher analysis for various cytokines.

Any adverse events experienced during this study will be documented.

ELIGIBILITY:
Inclusion Criteria:

* General good health
* Willing to adhere to the requirements of the protocol, including availability for follow-up visits
* Willing and able to sign written informed consent

Exclusion Criteria:

* Individuals with known HIV infection
* Individuals with malignancy
* Individuals with a history or symptoms of unstable cardiovascular disease
* Individuals with renal abnormalities
* Individuals having a history or symptoms of pulmonary disease
* Individuals having acute or active chronic liver disease
* Individuals having neurologic or psychiatric disease
* Individuals having active tuberculosis
* Individuals having multiple sclerosis
* Individuals having bleeding disorders
* Individuals with planned surgery over the course of the trial or having had major surgery in the past 6 mo.
* Individuals with a history of alcohol/drug abuse
* Pregnant and lactating women
* Individuals on prescribed medication with the exception of oral contraceptives
* Individuals with Crohn's disease, Lupus, Rheumatoid arthritis, Colitis or any other auto-immune disease
* Individuals using natural health products or dietary supplements for 2 weeks prior and during the trial
* Individuals having allergies to ginseng or to any known component of the drug product or placebo
* Smokers (smoking > 10 cigarettes/day)
* Alcoholics (drinking > 10 drinks/week)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-03; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
The change in innate and Th1 immune responses of the subjects

SECONDARY OUTCOMES:
Proportions of different leukocytes and lymphocytes in blood
Intracellular and plasma concentrations of various cytokines and immunoglobulins
Incidence and severity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Steven Sperber, MD, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hackensack University Medical Center, Hackensack, New Jersey, United States